CLINICAL TRIAL: NCT07291817
Title: Intermittent Negative Pressure for Patients With Diabetic Foot Ulcers (INPRESS) Study
Acronym: INPRESS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lo Zhiwen Joseph (Other Government)
Collaborators: Otivio AS (Industry)
Responsible Party: Sponsor-Investigator, Lo Zhiwen Joseph, Senior Consultant, Woodlands Health Campus
Organization: Woodlands Health Campus (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024-4641
Record Dates: First submitted 2025-11-16; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-11

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment with FlowOx (Experimental)
  Interventions: Device: FlowOx

INTERVENTIONS:
Device: FlowOx — 12 weeks treatment with FlowOx for 1 hour twice daily for 12 weeks

SUMMARY:
The aim of this trial is to investigate the safety and efficacy of 12 weeks treatment with FlowOx, for 1 hour twice daily, when used on patients with diabetic foot ulcers. The main question it aims to answer is whether treatment with FlowOx one hour in the morning and one hour in the evening for 12 weeks can improve toe arterial pressure and wound surface area compared to baseline.

Participants will have baseline assessments (i.e. toe pressure measurement and wound area measurement) performed on them and training on the use of FlowOx device will be provided to them in Visit 1. Participants will be tasked to use the FlowOx device (device will be loaned to them) for 1 hour twice daily. A phone call will be conducted 1 week after Visit 1 to follow up on the medical and user-related issues. At Week 6 (Visit 2), participants will be asked to come back for toe pressure and wound area measurement. At Week 12 (Visit 3), end of treatment assessments (i.e toe pressure and wound area measurement) will be performed. Compliance data will be acquired from the FlowOx device.

Their participation in the study will last for 12 weeks. Participants will be asked to use the FlowOx device for one hour, two times a day throughout the study period. They will need to visit the clinic 3 times in the course of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 21-99.
4. Diagnosed with diabetes mellitus.
5. Toe systolic pressure <70 mmHg on the leg to be treated (after revascularization)
6. Open chronic wound on the foot
7. Ability to operate the treatment device, and willing to adhere to the study intervention regimen.
8. Suitable for diabetic limb salvage

Exclusion Criteria:

1. Known allergic reactions to components of the INP device.
2. Treatment with another investigational intervention within the last 12 weeks prior to inclusion.
3. Pregnant women or cognitively impaired participants.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2026-11-02 (Estimated); Study Completion 2026-11-02 (Estimated)

PRIMARY OUTCOMES:
Change in toe arterial pressure | 12 weeks
  Toe systolic blood pressure is a commonly used tool to predict wound healing in patients with diabetic foot ulcers.
  * Tools used: Photoplethysmography (PPG) Probe/Sensor
  * Unit of measure: mmHg
Change in wound surface area | 12 weeks
  Change in wound surface area will be used as an indicator of treatment effect on wound healing.
  * Tool used: quantitative measurement of wound surface area
  * Unit of measure: cm2

SECONDARY OUTCOMES:
Comparison of the primary outcomes (changes in toe arterial pressure and wound healing rate) and post diabetic limb salvage rate between a prospective cohort that is 1:1 propensity-scored matched against a retrospective cohort | 12 weeks
  The prospective cohort will be 1:1 propensity-scored matched for age, gender and WIfI [wound, ischaemia, foot infection] score on presentation against a retrospective cohort.
  Post diabetic limb salvage rate:
  * Tools used: Rate of patients who do not undergo major LEA
  * Unit of measure: 12-week limb salvage rate
Frequency of adverse events | 12 weeks
  Adverse events and side effects of the treatment will be registered, so that safety assessments can be done during and after the trial.
Compliance (mean daily treatment time) | 12 weeks
  Compliance will be recorded as mean daily treatment time (registered by the device), so that exploratory sub-group analyses on patients with a certain compliance level may be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiwen Joseph Lo, Principal Investigator — Woodlands Health
Locations (1):
- Woodlands Health, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
IPD will be made available on a data repository if required by the publishing journal.

REFERENCES:
- [Background] Yagshyyev S, Hausmann P, Li Y, Kempf J, Zetzmann K, Dessi K, Moosmann O, Almasi-Sperling V, Meyer A, Gerken ALH, Lang W, Rother U. Intermittent negative pressure therapy in patients with no-option chronic limb-threatening ischemia. Vasa. 2023 Nov;52(6):402-408. doi: 10.1024/0301-1526/a001098. Epub 2023 Oct 17. PMID 37847243
- [Background] Herrmann LG, Reid MR. THE CONSERVATIVE TREATMENT OF ARTERIOSCLEROTIC PERIPHERAL VASCULAR DISEASES: PASSIVE VASCULAR EXERCISES (PAVAEX THERAPY). Ann Surg. 1934 Oct;100(4):750-60. doi: 10.1097/00000658-193410000-00016. No abstract available. PMID 17856393
- [Background] Landis E.M HLH. The clinical value of alternate suction and pressure in the treatment of advanced peripheral vascular disease. The American Journal of the Medical Sciences. 1935;189(3):20.
- [Background] Sinkowitz S, Gottlieb I. Thrombo-angiitis obliterans the conservative treatment by Bier's hyperemia suction apparatus. JAMA.1917;LXVIII(13):961-963.
- [Background] Sundby OH, Hoiseth LO, Mathiesen I, Jorgensen JJ, Sundhagen JO, Hisdal J. The effects of intermittent negative pressure on the lower extremities' peripheral circulation and wound healing in four patients with lower limb ischemia and hard-to-heal leg ulcers: a case report. Physiol Rep. 2016 Oct;4(20):e12998. doi: 10.14814/phy2.12998. PMID 27798353
- [Background] Sundby OH, Irgens I, Hoiseth LO, Mathiesen I, Lundgaard E, Haugland H, Weedon-Fekjaer H, Sundhagen JO, Sandbaek G, Hisdal J. Intermittent mild negative pressure applied to the lower limb in patients with spinal cord injury and chronic lower limb ulcers: a crossover pilot study. Spinal Cord. 2018 Apr;56(4):372-381. doi: 10.1038/s41393-018-0080-4. Epub 2018 Mar 1. PMID 29497177
- [Background] Hoel H, Pettersen EM, Hoiseth LO, Mathiesen I, Seternes A, Hisdal J. A randomized controlled trial of treatment with intermittent negative pressure for intermittent claudication. J Vasc Surg. 2021 May;73(5):1750-1758.e1. doi: 10.1016/j.jvs.2020.10.024. Epub 2020 Oct 22. PMID 33899743
- [Background] Sundby OH, Hoiseth LO, Mathiesen I, Weedon-Fekjaer H, Sundhagen JO, Hisdal J. The acute effects of lower limb intermittent negative pressure on foot macro- and microcirculation in patients with peripheral arterial disease. PLoS One. 2017 Jun 7;12(6):e0179001. doi: 10.1371/journal.pone.0179001. eCollection 2017. PMID 28591174
- [Background] Hoel H, Hoiseth LO, Sandbaek G, Sundhagen JO, Mathiesen I, Hisdal J. The acute effects of different levels of intermittent negative pressure on peripheral circulation in patients with peripheral artery disease. Physiol Rep. 2019 Oct;7(20):e14241. doi: 10.14814/phy2.14241. PMID 31631579
- [Background] Prompers L, Huijberts M, Apelqvist J, Jude E, Piaggesi A, Bakker K, Edmonds M, Holstein P, Jirkovska A, Mauricio D, Ragnarson Tennvall G, Reike H, Spraul M, Uccioli L, Urbancic V, Van Acker K, van Baal J, van Merode F, Schaper N. High prevalence of ischaemia, infection and serious comorbidity in patients with diabetic foot disease in Europe. Baseline results from the Eurodiale study. Diabetologia. 2007 Jan;50(1):18-25. doi: 10.1007/s00125-006-0491-1. Epub 2006 Nov 9. PMID 17093942
- [Background] Petersen BJ, Linde-Zwirble WT, Tan TW, Rothenberg GM, Salgado SJ, Bloom JD, Armstrong DG. Higher rates of all-cause mortality and resource utilization during episodes-of-care for diabetic foot ulceration. Diabetes Res Clin Pract. 2022 Feb;184:109182. doi: 10.1016/j.diabres.2021.109182. Epub 2022 Jan 18. PMID 35063288
- [Background] Armstrong DG, Boulton AJM, Bus SA. Diabetic Foot Ulcers and Their Recurrence. N Engl J Med. 2017 Jun 15;376(24):2367-2375. doi: 10.1056/NEJMra1615439. No abstract available. PMID 28614678
- [Background] Zhang Y, Lazzarini PA, McPhail SM, van Netten JJ, Armstrong DG, Pacella RE. Global Disability Burdens of Diabetes-Related Lower-Extremity Complications in 1990 and 2016. Diabetes Care. 2020 May;43(5):964-974. doi: 10.2337/dc19-1614. Epub 2020 Mar 5. PMID 32139380